CLINICAL TRIAL: NCT00905190
Title: Single Dose Crossover Comparative Bioavailability Study To Assess the Effect of Food on the Pharmacokinetics of Ondansetron Modified-Release Capsules (EUR1025) in Healthy Male and Female Volunteers
Brief Title: Bioavailability Study of Anti Nausea Medication With and Without Food
Acronym: EUR-1025
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ODO-P8-689
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Nausea
MeSH Terms: conditions — Nausea | interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fed (Experimental): A single oral dose of ondansetron (1 x 24 mg) will be administered with approximately 240 ml of water in the morning. The ondansetron dose will be administered after a 10-hour overnight fast and thirty minutes after consuming a high-fat, high-caloric breakfast
  Interventions: Drug: Ondansetron
- Fasting (Experimental): A single oral dose of ondansetron (1 x 24 mg) will be administered with approximately 240 ml of water in the morning after a 10-hour overnight fast.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — 24 mg one time
  Other Names: EUR-1025

SUMMARY:
This study is to assess the effect of food on a single dose of EUR-1025 when taken with a meal and taken on an empty stomach.

DETAILED DESCRIPTION:
The objective of this study is to assess the effect of food on the pharmacokinetics of a single 24 mg dose of EUR-1025 administered as a novel modified-release capsule formulation under fed and fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers,
* Non- or ex-smokers,
* Of at least 21 years of age but not older than 55 years with a body mass index targeted to be at least 18.5 and less than 30 kg/m2,
* Healthy, normal lab values,
* Negative HIV, Hepatitis B & C and a negative ethyl alcohol and drug screen,
* Normal 12 lead ECG, negative human chorionic gonadotropin (hCG) for females.

Exclusion Criteria:

* No known hypersensitivity to Ondansetron or any related products,
* Presence of significant gastrointestinal, liver or kidney disease,or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects,
* History of significant gastrointestinal, liver or kidney disease,
* Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease,
* Suicidal tendency,
* History of or disposition to seizures, state of confusion, clinically relevant psychiatric disease,
* Presence of significant heart disease or disorder discovered on screening ECG,
* Females who are found to have a positive serum pregnancy test at screening or are nursing,
* Females of childbearing potential who refuse to use an acceptable contraceptive regimen from the screening visit and throughout the study,
* Maintenance therapy with any drug,
* Significant history of drug dependency or alcohol abuse (> 2 units of alcohol per day, intake of excessive alcohol, acute or chronic),
* Any clinically significant illness in the previous 28 days before day 1 of the study,
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin,fluconazole, ketoconazole,diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin and rifampin), in the previous 28 days before day 1 of this study,
* Volunteers who took an Investigational Product (in another clinical trial) or donated 50 ml or more of blood in the previous 28 days before day 1 of this study,
* Poor motivation, intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with the protocol requirements or inability to cooperate adequately,
* Inability to understand and to observe the instructions of the physician,
* Donation of 500 ml or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies) in the previous 56 days before day 1 of this study,
* Positive urine screening of drugs or abuse,
* Any history of tuberculosis and/or prophylaxis for tuberculosis,
* Positive results to HIV, HBsAg, or anti-HCV tests,
* No subjects will be allowed to enroll in this study more than once.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Effects of food on the pharmacokinetics of a single 24 mg dose of ondansetron administered under fed and fasting conditions | 1 dose on two separate days

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, M.D., Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma INc., Mount Royal, Quebec, Canada